CLINICAL TRIAL: NCT01713907
Title: Evaluation of the Ulthera® System for Obtaining Lift and Tightening of the Facial Tissue and Improvement in Jawline Definition and Submental Skin Laxity
Brief Title: Evaluation of the Ulthera® System for Treatment of the Face and Neck
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate study staff to appropriately manage trial.
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ULT-109
Record Dates: First submitted 2012-10-15; First posted 2012-10-25 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2013-02

CONDITIONS: Wrinkles; Rhytids; Skin Laxity
Keywords: Ultherapy™ treatment; Ulthera® System; Ulthera, Inc.; Ultrasound treatment for skin tightening
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ulthera® treatment (Experimental): All enrolled subjects will receive one full face and neck Ulthera® treatment.
  Interventions: Device: Ulthera® Treatment

INTERVENTIONS:
Device: Ulthera® Treatment — Focused ultrasound energy delivered below the surface of the skin.
  Other Names: Ultherapy™ System; Ulthera, Inc.

SUMMARY:
Up to 15 subjects will be enrolled. Enrolled subjects will receive one Ulthera® treatment on the face and neck. Follow-up visits will occur at 45, 90 and 180 days post-treatment. Study images will be obtained pre-treatment, immediately post-treatment, and at each follow-up visit.

DETAILED DESCRIPTION:
This is a prospective, single-center, pilot clinical trial to evaluate the efficacy of the Ulthera® System to improve jawline definition and submental skin laxity. Changes from baseline in the Fitzpatrick Facial Wrinkle Scale and facial pigmentation will be assessed at study follow-up visits. Global Aesthetic Improvement Scale scores, patient satisfaction questionnaires, and quality of life questionnaires will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 30 to 65 years.
* Subject in good health.
* Score of 1 to 6 on the Fitzpatrick's Classification of Wrinkling Scale.
* Mild to moderate rhytids in the periorbital or perioral region.
* Mild to moderate laxity in the areas to be treated, which includes length and depth of lines.
* Mild to moderate vertical perioral lines
* Mild to moderate marionette lines.
* Subjects who desire lift and tightening of periorbital, perioral, and cheek tissue, improvement in jawline definition and/or submental skin laxity
* Understands and accepts the obligation not to undergo any other procedures in the areas to be treated through the follow-up period.
* Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.

Exclusion Criteria:

* Presence of an active systemic or local skin disease that may affect wound healing.
* Severe solar elastosis.
* Excessive subcutaneous fat on the cheek.
* Excessive skin laxity on the lower face and neck.
* Deep wrinkles, numerous lines, with or without redundant skin in the areas to be treated.
* Excessive hooding with or without redundant skin in the areas to be treated.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Improvement in facial wrinkles and lifting and tightening of skin | 90 days post-treatment
  Outcome measure determined based on a masked, qualitative assessment of standardized photographs at 90 days post-treatment compared to baseline

SECONDARY OUTCOMES:
Overall aesthetic improvement | Participants will be followed up to 180 days post-treatment
  Aesthetic improvement determined based on GAIS scores at follow-up, and the change in facial pigmentation and Fitzpatrick Facial Wrinkle Scale scores from baseline.
Overall patient satisfaction | 90 and 180 day post-treatment
  Determined based on Patient Satisfaction and Quality of Life questionnaire scores.

CONTACTS AND LOCATIONS:
Overall Officials: Hema Sundaram, MD, Principal Investigator — Dermatology, Cosmetic & Laser Surgery
Locations (1):
- Dermatology, Cosmetic & Laser Surgery, Rockville, Maryland, United States